CLINICAL TRIAL: NCT01298492
Title: A Multicenter Open-label Extension Study To Assess Long-term Safety Of PF-00547659 In Subjects With Crohn's Disease OPERA II
Brief Title: A Study To Monitor Long-Term Treatment With PF-00547659
Acronym: OPERA II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: A7281007; 2010-024638-48 (EudraCT Number)
Record Dates: First submitted 2011-01-26; First posted 2011-02-17 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Crohn's Disease
Keywords: Active Crohn's disease; Anti-TNF Refractory; Immunosuppressant Refractory
MeSH Terms: conditions — Crohn Disease | interventions — ontamalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-Label Treatment (Experimental): Subjects eligible for this study will have completed the 12 week double blind induction period in study A7281006 and will be stratified by responders or non responders based on change in CDAI in that study, without unblinding treatment assignment from study A7281006. Additionally, subjects who have completed study A7281008
  Interventions: Drug: PF-00547659

INTERVENTIONS:
Drug: PF-00547659 — 75 mg SC once monthly for 72 weeks. Subjects may escalate to 225 mg or de-escalate to 22.5 mg one time.

SUMMARY:
This study provides open-label drug to eligible patients who have completed a prior study of PF-00547659. The primary endpoint for this study is long-term safety.

DETAILED DESCRIPTION:
The rationale for conducting this open-label extension (OLE) study is primarily to evaluate long term safety of PF 00547659. This protocol also provides the opportunity for continued treatment for subjects responding to treatment from the feeder study. It also provides an opportunity for initial treatment for subjects randomized to placebo in the feeder study. This is a multi center Phase 2, open label, safety extension study for feeder studies which evaluate PF 00546759 in subjects with moderate to severe Crohn's disease. Subjects eligible for this study will have completed the 12 week double blind induction period in study A7281006 and will be stratified by responders or non responders based on change in CDAI in that study, without unblinding treatment assignment from study A7281006. Additionally, subjects who have completed study A7281008 with a clinical response, as defined by that protocol, will also be eligible for this study and treated as "responders". All subjects entering this study must have discontinued immunosuppressant therapy.

Subjects entering this study will be given a 75 mg SC dose at baseline and then every 4 weeks through Week 72. After the active treatment period, the subjects will enter a 24 month follow up period including 6 monthly visits followed by 18 month extended contact (every 6 month telephone contacts). At Week 96, subjects will undergo an End of Study visit but will continue the every 6 month telephone contacts until Week 168.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 76 years of age.
* Subjects previously enrolled in study A7281006 who have completed the blinded 84 day (12 week) induction period or in study A7281008 who have completed Week 12 and have demonstrated a clinical response as defined by that protocol.

Exclusion Criteria:

* Subjects that have completed Day 84 (Week 12) of a PF-00547659 study but have experienced serious event(s) related to the investigational product, an unstable medical condition, or any other reason, in the opinion of the investigator, would hinder entry or participation in this study.
* Subjects who are taking any dose of azathioprine, 6-mercaptopurine or methotrexate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2016-07-27 (Actual); Study Completion 2016-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (111):
- United States (47):
  - UCSD Medical Center - Thorton Hospital, La Jolla, California
  - Community Clinical Trials, Orange, California
  - GastroDiagnostics, Orange, California
  - Clinical Research of the Rockies, Lafayette, Colorado
  - Rmga - Rmcr, Thornton, Colorado
  - Rocky Mountain Gastroenterology Associates, Thornton, Colorado
  - MGG Group Co., Inc., Washington D.C., District of Columbia
  - Florida Center for Gastroenterology, Largo, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Miami Crohn's and Colitis Center, Miami, Florida
  - University of Miami Hospital and Clinic (IP Shipment Only), Miami, Florida
  - University of Miami Hospital and Clinic, Miami, Florida
  - University of Miami Hospital, Miami, Florida
  - Citrus Ambulatory Surgery Center, Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Heartland Medical Research, Inc., Clive, Iowa
  - Iowa Digestive Disease Center, Clive, Iowa
  - Iowa Endoscopy Center (Colonoscopy Only), Clive, Iowa
  - Metropolitan Gastroenterology Group, PC - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - Center for Digestive Health, Troy, Michigan
  - Surgical Centers of Michigan, Troy, Michigan
  - Surgery Center of Columbia, Columbia, Missouri
  - Audrain Medical Center, Mexico, Missouri
  - Center for Digestive and Liver Diseases, Inc., Mexico, Missouri
  - Barnes-Jewish Hospital - Investigational Drug Services, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Center for Advanced Medicine, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - New York Hospital Queens, Flushing, New York
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - Nassau Gastroenterology Associates Office Based Surgery, Great Neck, New York
  - Nassau Gastroenterology Associates, P.C., Great Neck, New York
  - North Shore Primary Care, P.C., Great Neck, New York
  - Lenox Hill Endoscopy Center, New York, New York
  - Synergy First, New York, New York
  - Premier Medical Group of the Hudson Valley, PC, Poughkeepsie, New York
  - CTRC Hospital, UNC Memorial Hospital, Chapel Hill, North Carolina
  - North Carolina Memorial Hospital Endoscopy Center, Chapel Hill, North Carolina
  - UNC Hospitals, Chapel Hill, North Carolina
  - UNC Hospitals Endoscopy, Chapel Hill, North Carolina
  - Hillsborough Campus, Hillsborough, North Carolina
  - University of Washington Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Allegiance Research Specialists, Wauwatosa, Wisconsin
- Austria (2):
  - AKH Wien Universitaetsklinik fuer Innere Medizin III, Vienna
  - AKH Wien, Vienna
- Belgium (5):
  - Hospital Erasme, Brussels
  - UZ Gasthuisberg - Pharmacy, Leuven
  - UZ Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire De Liege-Domaine Universitaire du Sart Tilman, Liège
  - Centre Hospitalier de Mouscron, Mouscron
- Canada (2):
  - Oshawa Clinic, Oshawa, Ontario
  - Toronto Digestive Disease Associates Inc., Vaughan, Ontario
- France (8):
  - Hopital Beaujon, Clichy
  - CHRU de Lille, Pharamcie Centrale, Lille
  - CIC - Hopital Cardiologique, Lille
  - Hopital Huriez, CHRU de Lille, Lille
  - Hopital de l'Archet 2 - CHU de Nice, Nice
  - Hopital Saint-Louis, Paris
  - Hopital Nord, Saint-Priest-en-Jarez
  - Hopital Rangueil, Toulouse
- Germany (9):
  - Robert Bosch Krankenhaus GmbH, Stuttgart, Baden-Wurttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - "Charite - Campus Berlin Mitte Medizinische Klinik, Berlin
  - Charite, Universitaetsmedizin Berlin, Campus Virchow-Klinikum, Berlin
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH, Halle
  - Universitaetsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitaetsfrauenklinikum Schleswig-Holstein, Lübeck
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
  - Universitaetsklinik Regensburg, Regensburg
- Japan (6):
  - National Hospital Organization Takasaki General Medical Center, Takasaki, Gunma
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - The Jikei University Hospital, Minato-Ku, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - National Hospital Organization Hirosaki National Hospital, Aomori, Toyko
  - Chiba University Hospital, Chiba
- Netherlands (3):
  - Academic Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Maastricht University Medical Center, Maastricht
- Norway (4):
  - Sykehusapoteket Asker og Baerum, Gjettum, Norway
  - Oslo Universitetssykehus, Oslo
  - Lovisenberg Diakonale Sykehus, Oslo
  - Vestre Viken HF, Rud
- Poland (5):
  - Centrum Endoskopii Zabiegowej, Bydgoszcz
  - NZOZ Centrum Medyczne Szpital Sw. Rodziny, Lodz
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych i Administracji w Warszawie, Warsaw
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych W Warszawie, Warsaw
  - Lexmedica, Wroclaw
- Serbia (3):
  - Military Medical Academy, Belgrade
  - Clinical Hospital Centre Bezanijska Kosa, Belgrade
  - Clinical Hospital Center Zemun, Clinical Department for Gastroenterology and Hepatology, Zemun
- Slovakia (4):
  - Gastroentero-Hepatologicke centrum THALION, LAMA MEDICAL CARE s.r.o., Bratislava
  - Medak s.r.o., Bratislava
  - KM Management spol. s r.o., Nitra
  - Synergy group, a.s., Nové Mesto nad Váhom
- South Africa (3):
  - Wits Clinical Research, Johannesburg, Gauteng, South Africa
  - Parklands Medical Centre, Durban, KwaZulu-Natal
  - Kingsbury Hospital, Cape Town, Western Cape
- South Korea (5):
  - Yeungnam University Hospital, Daegu, Korea, Republic of
  - Pusan National University Hospital, Busan
  - Samsung Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (5):
  - Corporacio Sanitaria Parc Tauli de Sabadell, Sabadell, Barcelona
  - Corporacio Sanitaria Parc Tauli de Sabadell, Sabadell, Catalonia
  - Hospital Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid

REFERENCES:
- [Derived] D'Haens GR, Reinisch W, Lee SD, Tarabar D, Louis E, Klopocka M, Klaus J, Schreiber S, Il Park D, Hebuterne X, Nagy P, Cataldi F, Martin SW, Nayak S, Banerjee A, Gorelick KJ, Sandborn WJ. Long-Term Safety and Efficacy of the Anti-Mucosal Addressin Cell Adhesion Molecule-1 Monoclonal Antibody Ontamalimab (SHP647) for the Treatment of Crohn's Disease: The OPERA II Study. Inflamm Bowel Dis. 2022 Jul 1;28(7):1034-1044. doi: 10.1093/ibd/izab215. PMID 34427633
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7281007&StudyName=A%20Study%20To%20Monitor%20Long-Term%20Treatment%20With%20PF-00547659

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 81 centers in Austria, Belgium, Canada, France, Germany, Japan, Netherlands, Norway, Poland, Republic of Korea, Serbia, Slovakia, South Africa, Spain and United States between 22 July 2011 (first participant first visit) and 27 July 2016 (last participant last visit).
Pre-assignment Details: A total of 268 participants (225 participants from Feeder Study A7281006 [NCT01276509] and 43 participants from Feeder Study A7281008 [NCT01387594]) were enrolled and overall 149 participants completed the study.
Groups:
- PF-00547659 75 mg: Participants received PF-00547659 75 milligram (mg) subcutaneous injection once in every 4 weeks through Week 72. One time dose escalation to 225 mg subcutaneous injection was allowed after 8 weeks of the study for the participants who experienced clinical deterioration or unacceptably low level of response to study drug. One time dose de-escalation to 22.5 mg subcutaneous injection due to intolerance or AEs was also allowed after the investigator carefully assessed the status of the participant.
Period: Overall Study
Arm/Group | PF-00547659 75 mg
Started | 268
Completed | 149
Not Completed | 119
Not completed — Death | 2
Not completed — Insufficient Clinical Response | 22
Not completed — Lost to Follow-up | 12
Not completed — Withdrawal by Subject | 47
Not completed — Other (Unspecified) | 7
Not completed — Withdrawn Due to Pregnancy | 1
Not completed — Protocol Violation | 2
Not completed — Adverse Event(Related to Study Drug) | 8
Not completed — Adverse Event(Not Related to Study Drug) | 18

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (mITT) population included all enrolled participants who received at least 1 dose of investigational product.
Groups:
- PF-00547659 75 mg: Participants received PF-00547659 75 mg subcutaneous injection once in every 4 weeks through Week 72. One time dose escalation to 225 mg subcutaneous injection was allowed after 8 weeks of the study for the participants who experienced clinical deterioration or unacceptably low level of response to study drug. One time dose de-escalation to 22.5 mg subcutaneous injection due to intolerance or AEs was also allowed after the investigator carefully assessed the status of the participant.
Arm/Group | PF-00547659 75 mg
Number analyzed (Participants) | 268
Age, Continuous [Mean (Standard Deviation); unit: year] | 36.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151
  Male | 117

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With On-Treatment Adverse Events (AEs), AEs Led to Withdrawal, and Serious Adverse Events (SAEs)
Description: AEs included adverse drug reactions, illnesses with onset during the study, exacerbation of previous illnesses, clinically significant changes in physical examination findings and abnormal objective test findings (ECG, laboratory). An SAE was defined as any AE at any dose that resulted in death; was life threatening (immediate risk of death); required in-subject hospitalization or prolongation of existing hospitalization; resulted in a persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); or resulted in congenital anomaly/birth defect.
Time Frame: From start of study treatment up to Week 72 (Treatment Period)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PF-00547659 75 mg
Number analyzed (Participants) | 268
Participants
  Participants With AEs | 249
  Participants With AEs Led to Withdrawal | 53
  Participants With SAEs | 80

2. Secondary Outcome: Number of Participants With Positive Anti-Drug (PF-00547659) Antibodies
Description: Positive Anti-Drug Antibodies result was defined as ADA titre value greater than or equal to (>=) 4.64 at at least one of the time points.
Time Frame: Baseline up to Week 96
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PF-00547659 75 mg
Number analyzed (Participants) | 268
Participants | 63

3. Secondary Outcome: Serum Trough Concentrations of PF-00547659 Versus Time
Description: Serum trough concentrations of PF-00547659 were analyzed using population Pharmacokinetic (PK) methodology.
Time Frame: Week 4,8,12,16,20,24,28,32,36,40,44,48,52,56,60,64,68,72,76,80,84,88,92,96
Population: PK population included all enrolled participants who received at least 1 dose of investigational product and had data on at least 1 PK concentration.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-00547659 75 mg
Number analyzed (Participants) | 260
nanogram per milliliter (ng/mL)
  Week 4: number analyzed (Participants) | 226
  Week 4 | 6673 (6634.2)
  Week 8: number analyzed (Participants) | 222
  Week 8 | 6064 (4455.3)
  Week 12: number analyzed (Participants) | 201
  Week 12 | 8040 (6293.1)
  Week 16: number analyzed (Participants) | 188
  Week 16 | 9563 (7285.4)
  Week 20: number analyzed (Participants) | 186
  Week 20 | 10400 (8438.6)
  Week 24: number analyzed (Participants) | 172
  Week 24 | 10450 (7934.6)
  Week 28: number analyzed (Participants) | 162
  Week 28 | 10780 (9211.0)
  Week 32: number analyzed (Participants) | 165
  Week 32 | 11920 (10675)
  Week 36: number analyzed (Participants) | 164
  Week 36 | 12460 (9717.1)
  Week 40: number analyzed (Participants) | 152
  Week 40 | 12570 (10077)
  Week 44: number analyzed (Participants) | 149
  Week 44 | 12960 (10999)
  Week 48: number analyzed (Participants) | 148
  Week 48 | 13170 (11108)
  Week 52: number analyzed (Participants) | 144
  Week 52 | 13560 (11388)
  Week 56: number analyzed (Participants) | 134
  Week 56 | 13930 (11191)
  Week 60: number analyzed (Participants) | 131
  Week 60 | 14130 (11095)
  Week 64: number analyzed (Participants) | 127
  Week 64 | 14360 (11290)
  Week 68: number analyzed (Participants) | 120
  Week 68 | 14990 (12883)
  Week 72: number analyzed (Participants) | 114
  Week 72 | 13910 (10554)
  Week 76: number analyzed (Participants) | 173
  Week 76 | 10520 (10082)
  Week 80: number analyzed (Participants) | 170
  Week 80 | 3555 (5339.8)
  Week 84: number analyzed (Participants) | 149
  Week 84 | 1129 (2634.7)
  Week 88: number analyzed (Participants) | 145
  Week 88 | 403.8 (1522.6)
  Week 92: number analyzed (Participants) | 136
  Week 92 | 154.2 (1001.9)
  Week 96: number analyzed (Participants) | 145
  Week 96 | 54.73 (487.07)

ADVERSE EVENTS:
Time Frame: From Start of Study Treatment up to Safety Follow up (Week 96)
Arm/Group | PF-00547659 75 mg
All-Cause Mortality (participants affected / at risk) | 2/268
Serious Adverse Events (participants affected / at risk) | 118/268
Other Adverse Events (participants affected / at risk) | 206/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-00547659 75 mg (N=268)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis enteropathic (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Anal fistula (Gastrointestinal disorders) | 7 (7)
Anal stenosis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 44 (51)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 4 (4)
Intestinal fistula (Gastrointestinal disorders) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (4)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (11)
Vomiting (Gastrointestinal disorders) | 3 (3)
General physical health deterioration (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (3)
Coronary artery disease (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 2 (2)
Abdominal wall abscess (Infections and infestations) | 2 (2)
Abscess intestinal (Infections and infestations) | 1 (1)
Abscess neck (Infections and infestations) | 1 (1)
Anal abscess (Infections and infestations) | 10 (10)
Clostridium difficile infection (Infections and infestations) | 3 (3)
Device related infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1)
Pelvic abscess (Infections and infestations) | 2 (2)
Perirectal abscess (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 4 (5)
Postoperative abscess (Infections and infestations) | 1 (1)
Rotavirus infection (Infections and infestations) | 1 (1)
Splenic abscess (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Vulval abscess (Infections and infestations) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (3)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Stomal hernia (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Blood creatine phosphokinase mm increased (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1)
Bladder dysfunction (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Ureterolithiasis (Renal and urinary disorders) | 1 (1)
Urinoma (Renal and urinary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Hepatic cyst (Hepatobiliary disorders) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 (1)
Benign breast lump removal (Surgical and medical procedures) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Perineal fistula (Reproductive system and breast disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-00547659 75 mg (N=268)
Arthralgia (Musculoskeletal and connective tissue disorders) | 83 (113)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (30)
Abdominal pain (Gastrointestinal disorders) | 49 (59)
Anal fissure (Gastrointestinal disorders) | 14 (14)
Aphthous ulcer (Gastrointestinal disorders) | 14 (18)
Crohn's disease (Gastrointestinal disorders) | 79 (111)
Diarrhoea (Gastrointestinal disorders) | 24 (38)
Nausea (Gastrointestinal disorders) | 32 (44)
Vomiting (Gastrointestinal disorders) | 23 (34)
Asthenia (General disorders) | 15 (20)
Fatigue (General disorders) | 20 (23)
Pyrexia (General disorders) | 27 (36)
Anal abscess (Infections and infestations) | 14 (16)
Bronchitis (Infections and infestations) | 20 (26)
Gastroenteritis (Infections and infestations) | 19 (22)
Influenza (Infections and infestations) | 18 (19)
Nasopharyngitis (Infections and infestations) | 54 (93)
Pharyngitis (Infections and infestations) | 15 (18)
Upper respiratory tract infection (Infections and infestations) | 20 (25)
Urinary tract infection (Infections and infestations) | 19 (28)
Headache (Nervous system disorders) | 35 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right to review disclosures, requesting a delay of up to 60 days. The first publication must be a joint publication covering all centers. However, if a joint manuscript has not been submitted for publication within 12 months of completion or termination of study at all participating sites, Investigator may publish individual site results separately. Investigator may not disclose previously undisclosed confidential information other than study results.